CLINICAL TRIAL: NCT06236100
Title: Evaluating an Adverse Childhood Experience-Targeting Advocate Model of a Substance Use Prevention Program: A Hybrid Type 1 Effectiveness-Implementation Trial
Brief Title: Evaluating an Adverse Childhood Experience-Targeting Advocate Model of a Substance Use Prevention Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: New Jersey Prevention Network (Unknown); RWJBarnabas Health Institute for Prevention and Recovery (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0218779
Record Dates: First submitted 2023-12-26; First posted 2024-02-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Substance-Related Disorders; Adverse Childhood Experiences
Keywords: Adverse Childhood Experiences; Strengthening Families Program; Family Advocate; Community-level interventions; Hybrid Type 1 Design; Mixed-Method Evaluation; Effectiveness Trial; Cluster Randomized Controlled Trial; Process Evaluation; Cost Evaluation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening Families Program + Family Advocate (Experimental): Families in the treatment group will be connected to clinically trained, trauma-informed FAs that will assess and refer families to community services. The intervention will provide wraparound supports to prevent ACEs and substance use and, critically, enable providers and community-based partners to align their services in a way that addresses the social determinants of health and other community-level factors that impact substance use and the relationship between social connection and ACEs. The FA component of the intervention will run concurrent to the Strengthening Families Program 7-17 sessions, with the FAs interacting weekly with families over the 10- to 14-week intervention period. On a weekly basis, FAs will conduct 1-hour, post-session check-ins with each family. This 1-hour period will consist of a 20-minute phone call with families to discuss their needs, with the remaining 40 minutes used to debrief, make service referrals, and complete documentation.
  Interventions: Behavioral: Strengthening Families Program + Family Advocate
- Strengthening Families Program-Only (Active Comparator): Families in the control group will participate in the Strengthening Families Program 7-17 (SFP7-17) Group Class Curriculum for families with children ages 7-17. Parents and children participate in SFP7-17, both separately and together, as the curriculum has lessons for parents, teens, and children plus a joint Family Practice class. SFP7-17 meetings are 2 hours in length and are typically held in person (but families can participate remotely, during extenuating circumstances) with participating families completing 11 sessions over a 10- to 14-week period.
  Interventions: Behavioral: Strengthening Families Program

INTERVENTIONS:
Behavioral: Strengthening Families Program + Family Advocate — This intervention will integrate clinically trained, trauma-informed Family Advocates (FA) into the established, evidence-based Strengthening Families Program (SFP). Families will participate in the SFP7-17 curriculum, which consists of 11 sessions over 10-14 weeks. FAs will assist families in accessing community resources for substance use and Adverse Childhood Experiences (ACE) prevention and treatment.
  Arms: Strengthening Families Program + Family Advocate
Behavioral: Strengthening Families Program — This intervention consists of the SFP7-17 Group Class Curriculum. Families will participate in the SFP7-17 curriculum, which consists of 11 sessions over 10-14 weeks.
  Arms: Strengthening Families Program-Only

SUMMARY:
Primary Objective: Conduct a rigorous evaluation of a prevention-based intervention designed to mitigate the harms of adverse childhood experiences (ACEs) exposure and prevent future ACEs, substance use, and overdose within 36 communities experiencing a disproportionate burden of substance use and ACEs.

The study has three aims: (1) use a cluster randomized controlled trial to test effectiveness of the Strengthening Families Program (SFP) + Family Advocate (FA) intervention on substance use, overdose, and ACEs in 18 communities compared with SFP-only in 18 communities; (2) conduct a robust process evaluation informed by the Consolidated Framework for Implementation Research (CFIR) to explore implementation barriers and facilitators; and (3) conduct a cost evaluation to accurately estimate the costs required to implement SFP and SFP+FA and assess the cost-effectiveness of SFP+FA relative to SFP alone. Findings will provide a roadmap about the best ways to help disproportionately affected communities prevent substance use, overdose, and ACEs.

DETAILED DESCRIPTION:
Early exposure to Adverse Childhood Experiences (ACEs), such as parental substance use, increases the likelihood of future substance use and drug overdose, resulting in an intergenerational cycle of substance-related ACEs that can continue indefinitely if left uninterrupted. Community-level interventions may moderate the relationship between ACEs and substance use by providing an array of family support services and treatments to reduce disparities and improve reach and service linkages in the community. Although research suggests that effectively decreasing the prevalence and impact of ACEs and substance use requires addressing both family- and community-level factors in tandem, there is a critical gap within the evidence base pertaining to interventions that effectively integrate the two factors to prevent substance use and ACEs. RTI International and its partners, the New Jersey Prevention Network and RWJBarnabas Health, will evaluate an intervention integrating New Jersey's established, evidence-based Strengthening Families Program (SFP) with clinically trained, trauma-informed Family Advocates (FAs) who will assist families (i.e., parents/caregivers and youth between the ages of 12 and17) in accessing community resources. Specifically, this study will use a Hybrid Type 1 effectiveness-implementation design across 36 New Jersey communities experiencing a disproportionate burden of substance use and ACEs.

ELIGIBILITY:
Inclusion Criteria: To be eligible to participate in this study, a family must meet all of the following criteria:

* Either reside in, or attend SFP meetings, within one of the 36 New Jersey communities with disproportionate levels of ACEs and substance use disorder (SUD) issues that are assigned to either the treatment or control conditions via the study's cluster randomized controlled trial design
* Meet family eligibility requirements:

  * One or more adult caregivers
  * One or more adolescents, ages 7 to 17
* Caregiver provision of signed and dated informed consent form
* For children, informed assent and parental permission via the informed consent to participate in the study
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Willingness to adhere to the regimens of the SFP and FA interventions
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, smart phone, internet access)

Exclusion Criteria: A family who meets any of the following criteria will be excluded from participation in this study:

* Caregiver has previously completed SFP with one or more children, ages 7 to 17
* Intellectual disabilities (i.e., cognitive impairments that would prohibit the completion of the SFP curriculum or data collection instruments)
* Language difficulties (caregivers and children must read and understand spoken English)

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Substance use prevalence | Baseline, intervention completion (ranging from 10 to 14 weeks), and 6-month post-intervention follow-up
  Measure of substance use prevalence among parents/caregivers and youth derived from 4 questions included on the SFP adult and SFP youth pre-test, post-test, and 6-month follow-up surveys. These 4 questions focus on whether various substances were ever used, used in the past 30 days, on how many day substances were used (if any), and which substances were used.
Substance use perceptions of harm | Baseline, intervention completion (ranging from 10 to 14 weeks), and 6-month post-intervention follow-up
  Measure of substance use perceptions of harm among parents/caregivers and youth derived from 3 questions included on the SFP adult and SFP youth pre-test, post-test, and 6-month follow-up surveys. These 3 questions focus on perceptions of harm associated with alcoholic beverages, marijuana, and prescription drugs.
Referrals to clinical services | Baseline, intervention completion (ranging from 10 to 14 weeks), and 6-month post-intervention follow-up
  Measure of rate of referrals to clinical services among participating families using the study's Weekly Clinical and Non-Clinical Services Referral Log
Referrals to non-clinical services | Baseline, intervention completion (ranging from 10 to 14 weeks), and 6-month post-intervention follow-up
  Measure of rate of referrals to non-clinical services among participating families using the study's Weekly Clinical and Non-Clinical Services Referral Log

SECONDARY OUTCOMES:
ACEs prevalence | Baseline and 6-month post-intervention follow-up
  Measure of ACEs prevalence among parents/caregivers and youth in participating families using 3 questions from the study's pre-test and 6-month post-test ACEs/Social Needs Screener. These 3 questions focus on the prevalence of the three main ACEs categories of abuse, neglect, and household challenges.
Social needs prevalence | Baseline and 6-month post-intervention follow-up
  Measure of social needs prevalence among parents/caregivers and youth in participating families using 18 questions from the study's pre-test and 6-month post-test ACEs/Social Needs Screener. These 18 questions correspond to 5 social determinants of health domains (including house, food security, transportation, finances, and personal safety) from the American Academy of Family Physicians' social determinants of health screening tool.
Substance use risk | Baseline, intervention completion (ranging from 10 to 14 weeks), and 6-month post-intervention follow-up
  Measure of substance use risk among parents/caregivers and youth derived from 3 questions included on the SFP adult and SFP youth pre-test, post-test, and 6-month follow-up surveys. These 3 questions focus on ease of access to different types of substances that may increase risk of substance use.
System linkages | Baseline and 6-month post-intervention follow-up
  Measures of change in clinical and non-clinical referral networks (such as changes in network size, edges, density, centrality, reciprocity, triadic closure, and assortativity) using questions included on the study's pre-test and 6-month post-test community service provider survey
Average start-up cost | Pre-implementation
  Measure of average cost per agency of starting up a program to deliver the intervention or active comparator using data from the study's Costing Instrument and Interview and administrative data from the New Jersey Prevention Network
Intervention cost | Intervention start to intervention completion (ranging from 10 to 14 weeks)
  Measure of intervention cost at the participant level of delivering the intervention or active comparator using data from the study's Costing Instrument and Interview, 4 questions from the Intervention Cost Survey for SFP Facilitators, and 2 questions from the Intervention Cost Survey for Family Advocates
Cost per service referral | Intervention start to intervention completion (ranging from 10 to 14 weeks)
  Measure of cost per service referral at the participant level using data from outcomes 6, 7, and 12, comparing cost per service referral for treatment and active comparator

OTHER OUTCOMES:
Service utilization | Baseline and 6-month post-intervention follow-up
  Referred service utilization rates among participating families in the treatment and active comparator using data from the SFP adult and SFP youth post-test, and 6-month follow-up surveys
Treatment/service adherence | Baseline and 6-month post-intervention follow-up
  Referred treatment/service adherence rates among participating families in the treatment and active comparator using data from the SFP adult and SFP youth post-test, and 6-month follow-up surveys
Lessons learned (process evaluation) | Pre-implementation to intervention completion (ranging from 10 to 14 weeks)
  Lessons learned related to implementing the intervention using data from the Post-Trial Focus Groups and Prevention Agency Program Lead Interviews
Social connectedness across systems (process evaluation) | Pre-implementation to intervention completion (ranging from 10 to 14 weeks)
  Extent that implementation of the intervention facilitates increased cross-system coordination and communication among the agencies that support families using data from the Post-Trial Focus Groups and Prevention Agency Program Lead Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Phillip W. Graham, DrPH, Principal Investigator — RTI International; Dallas J Elgin, PhD, Principal Investigator — RTI International
Locations (1):
- New Jersey Prevention Network, Tinton Falls, New Jersey, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT06236100/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT06236100/ICF_001.pdf